CLINICAL TRIAL: NCT02831829
Title: Comparative Effect of Water-based and Land-based Exercise Training on Exercise Capacity and Other Selected Cardiovascular Parameters in Patients With Coronary Artery Disease
Brief Title: Influence of Different Forms of Exercise Training in Patients With Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: KRKA (Industry)
Responsible Party: Principal Investigator, Borut Jug, Assistant professor, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKCLRehab0012016
Record Dates: First submitted 2016-07-11; First posted 2016-07-13 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Coronary Artery Disease
Keywords: cardiac rehabilitation; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Water-based exercise training group (Active Comparator): Intervention: Patients randomized to the "water-based exercise training group" will undergo water-based exercise training. The immersed exercise will include two session of aerobic (water-based) and calisthenic exercise per day, six days of a week, each lasting 30 minutes.
  Interventions: Other: water-based exercise training
- Land-based exercise training group (Active Comparator): Patients randomized to the "land-based exercise training group" will undergo exercise training which will include two aerobic and calisthenic exercise session per day, six days of a week, lasting 30 minutes
  Interventions: Other: land-based exercise training
- Control group (usual care) (No Intervention): Control group: patients randomized in control group will have usual care with no exercise

INTERVENTIONS:
Other: water-based exercise training — Water-based training will be performed in upright position, in waist to xyphoid process deep thermo-neutral water at temperature of 32,8 C. The immersed exercise will include two session of aerobic and calisthenic exercise per day, six days of a week, both lasting 30 minutes
  Arms: Water-based exercise training group
Other: land-based exercise training — Land-based training will include two aerobic and calisthenic exercise session per day, six days of a week, both lasting 30 minutes
  Arms: Land-based exercise training group

SUMMARY:
The aim of the study is to compare the effect of water-based and land-based exercise training, and usual care (no exercise training) in patient with coronary artery disease, on exercise capacity, vascular function, arrhythmogenic potential and cardiac autonomic function, and markers of neurohormonal activity, activated hemostasis and inflammation.

DETAILED DESCRIPTION:
Swimming and other water-based physical activities represent an effective form of aerobic-dynamic exercise. However, existing guidelines mainly advise caution when recommending water-based activities to patients with coronary artery disease. To date, safety and efficacy of short-term water-based exercise in patients with coronary artery diseases have only scarcely been addressed.

Cardiovascular rehabilitation is an integral part of management after a myocardial infarction or coronary procedure. Most rehabilitation programs are exercise-based, since the beneficial effects of physical activity undisputed, and corroborated by a large body of evidence.

Most rehabilitation programs are exercise-based, since the beneficial effects of physical activity undisputed, and corroborated by a large body of evidence.

Research has mainly been focused on the impact assessment of the standard forms of physical training, they studied various forms of physical exercise, mainly land-based. No previous study has reported on the effect of exercise in water as an integral element of standard cardiac rehabilitation in coronary patients on exercise capacity, vascular function, arrhythmogenic potential and cardiac autonomic function, and markers of neurohormonal activity, activated hemostasis and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* patients with coronary artery disease after myocardial infarction or myocardial revascularization (percutaneous coronary procedure or surgical revascularization)

Exclusion Criteria:

* unstable coronary artery disease, ejection fraction of the left ventricle of 40% or less, heart valve defect that dictate specific treatment, condition after valve replacement, heart rhythm disorders, the presence of a permanent pacemaker, contraindications to exercise, inability to perform exercise testing, mental retardation, severe anemia, obstructive/restrictive lung disease severe degree, recent thrombo embolic events, age over 80 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-05; Primary Completion 2016-10 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Change of maximal oxygen consumption during cardiopulmonary bicycle exercise testing | 14 days

SECONDARY OUTCOMES:
Change of flow-mediated dilation of brachial artery measured in % | 14 days
Change of arrhythmogenic potential estimated by high resolution ECG | 14 days
Change of the C-reactive protein serum concentration value, measured in g/l | 14 days
Change of N terminal - proBNP serum concentration value , measured in ng/l | 14 days
Change of the D-dimer serum concentration value, measured in microg/l | 14 days
Change in fibrinogen serum concentration value, measured in g/l | 14 days
Change of from-the-questionnaire-obtained quality of life, measured in points | 14 days
Change in heart rate variability, estimated by high resolution ECG | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Borut Jug, MD, PhD, Study Chair — University Medical Centre Ljubljana
Locations (2):
- Slovenia (2):
  - University medical center Ljubljana, Ljubljana
  - Terme Krka, Novo Mesto

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Piepoli MF, Corra U, Benzer W, Bjarnason-Wehrens B, Dendale P, Gaita D, McGee H, Mendes M, Niebauer J, Zwisler AD, Schmid JP; Cardiac Rehabilitation Section of the European Association of Cardiovascular Prevention and Rehabilitation. Secondary prevention through cardiac rehabilitation: from knowledge to implementation. A position paper from the Cardiac Rehabilitation Section of the European Association of Cardiovascular Prevention and Rehabilitation. Eur J Cardiovasc Prev Rehabil. 2010 Feb;17(1):1-17. doi: 10.1097/HJR.0b013e3283313592. PMID 19952757
- [Background] Aspry K, Wu WC, Salmoirago-Blotcher E. Cardiac Rehabilitation in Patients with Established Atherosclerotic Vascular Disease: New Directions in the Era of Value-Based Healthcare. Curr Atheroscler Rep. 2016 Feb;18(2):10. doi: 10.1007/s11883-016-0561-x. PMID 26803511
- [Background] St John Sutton M, Lee D, Rouleau JL, Goldman S, Plappert T, Braunwald E, Pfeffer MA. Left ventricular remodeling and ventricular arrhythmias after myocardial infarction. Circulation. 2003 May 27;107(20):2577-82. doi: 10.1161/01.CIR.0000070420.51787.A8. Epub 2003 May 5. PMID 12732606
- [Background] McDermott MM, Greenland P, Guralnik JM, Ferrucci L, Green D, Liu K, Criqui MH, Schneider JR, Chan C, Ridker P, Pearce WH, Martin G, Clark E, Taylor L. Inflammatory markers, D-dimer, pro-thrombotic factors, and physical activity levels in patients with peripheral arterial disease. Vasc Med. 2004 May;9(2):107-15. doi: 10.1191/1358863x04vm525oa. PMID 15521700
- [Background] Passino C, Severino S, Poletti R, Piepoli MF, Mammini C, Clerico A, Gabutti A, Nassi G, Emdin M. Aerobic training decreases B-type natriuretic peptide expression and adrenergic activation in patients with heart failure. J Am Coll Cardiol. 2006 May 2;47(9):1835-9. doi: 10.1016/j.jacc.2005.12.050. Epub 2006 Apr 19. PMID 16682309
- [Background] Swardfager W, Herrmann N, Cornish S, Mazereeuw G, Marzolini S, Sham L, Lanctot KL. Exercise intervention and inflammatory markers in coronary artery disease: a meta-analysis. Am Heart J. 2012 Apr;163(4):666-76.e1-3. doi: 10.1016/j.ahj.2011.12.017. PMID 22520533
- [Background] Autenrieth C, Schneider A, Doring A, Meisinger C, Herder C, Koenig W, Huber G, Thorand B. Association between different domains of physical activity and markers of inflammation. Med Sci Sports Exerc. 2009 Sep;41(9):1706-13. doi: 10.1249/MSS.0b013e3181a15512. PMID 19657301
- [Background] Hammett CJ, Prapavessis H, Baldi JC, Varo N, Schoenbeck U, Ameratunga R, French JK, White HD, Stewart RA. Effects of exercise training on 5 inflammatory markers associated with cardiovascular risk. Am Heart J. 2006 Feb;151(2):367.e7-367.e16. doi: 10.1016/j.ahj.2005.08.009. PMID 16442901
- [Background] Teffaha D, Mourot L, Vernochet P, Ounissi F, Regnard J, Monpere C, Dugue B. Relevance of water gymnastics in rehabilitation programs in patients with chronic heart failure or coronary artery disease with normal left ventricular function. J Card Fail. 2011 Aug;17(8):676-83. doi: 10.1016/j.cardfail.2011.04.008. Epub 2011 May 31. PMID 21807330
- [Background] Vona M, Codeluppi GM, Iannino T, Ferrari E, Bogousslavsky J, von Segesser LK. Effects of different types of exercise training followed by detraining on endothelium-dependent dilation in patients with recent myocardial infarction. Circulation. 2009 Mar 31;119(12):1601-8. doi: 10.1161/CIRCULATIONAHA.108.821736. Epub 2009 Mar 16. PMID 19289636
- [Background] Tokmakidis SP, Spassis AT, Volaklis KA. Training, detraining and retraining effects after a water-based exercise program in patients with coronary artery disease. Cardiology. 2008;111(4):257-64. doi: 10.1159/000127737. Epub 2008 Apr 23. PMID 18434735
- [Derived] Vasic D, Novakovic M, Bozic Mijovski M, Barbic Zagar B, Jug B. Short-Term Water- and Land-Based Exercise Training Comparably Improve Exercise Capacity and Vascular Function in Patients After a Recent Coronary Event: A Pilot Randomized Controlled Trial. Front Physiol. 2019 Jul 16;10:903. doi: 10.3389/fphys.2019.00903. eCollection 2019. PMID 31379605